CLINICAL TRIAL: NCT02049931
Title: The Comparative Study for Treatment Outcomes of Osteoporotic Compression Fracture Without Neurologic Injury Using Rigid Brace, Soft Brace, and no Brace
Brief Title: Comparison of Treatments of Osteoporotic Compression Fracture Using Rigid Brace, Soft Brace, and no Brace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Brace001
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Compression Fracture
Keywords: osteoporosis, compression fracture, brace
MeSH Terms: conditions — Fractures, Compression; Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No brace group (Experimental): Patients in the no brace treatment group were allowed to ambulate without any braces as long as it would be tolerable.
  Interventions: Device: No brace treatment
- Rigid brace group (Active Comparator): Patients in the rigid brace immobilization group were strictly maintained on bed rest until fitted a thoraco-lumbo-sacral orthosis. Brace is required to be worn at all times except when lying. All patients were instructed to wear the rigid brace for a total of 8 weeks.
  Interventions: Device: Rigid brace
- Soft brace group (Active Comparator): Because soft back brace was a custom-made, it began to be worn when enrollment for the study. Brace is required to be worn at all times except when lying. All patients were instructed to wear the soft brace for a total of 8 weeks.
  Interventions: Device: Soft brace

INTERVENTIONS:
Device: No brace treatment — Patients in the no brace group were allowed to ambulate without any braces as long as it would be tolerable.
  Arms: No brace group
Device: Rigid brace — In rigid brace group, brace is required to be worn at all times except when lying. All patients were instructed to wear the rigid brace for a total of 8 weeks.
  Arms: Rigid brace group
Device: Soft brace — In soft brace group, brace is required to be worn at all times except when lying. All patients were instructed to wear the soft brace for a total of 8 weeks.
  Arms: Soft brace group

SUMMARY:
The treatment outcomes in the treatment without brace would be non-inferior to those in use of rigid or soft brace.

DETAILED DESCRIPTION:
Bracing has been considered as a landmark step in conservative management for osteoporotic compression fractures. However, no prospective, randomized, and controlled clinical trials are available to document for the efficacy of wearing of the rigid or soft brace for the management of osteoporotic compression fracture. Therefore, the current trial was therefore designed to compare the outcome for improvement of disability and pain in patients with osteoporotic compression fracture using rigid, soft, or no brace.

ELIGIBILITY:
Inclusion Criteria:

* the presence of acute back pain caused by a single level vertebral fracture within 3 days of minor trauma such as fall from height,
* compression fracture between T 7 and L3 including injuries of only anterior compartment of vertebral body without neurologic deficit.

Exclusion Criteria:

* the presence of more than two recent vertebral fractures,
* pathologic malignant compression fractures,
* neurologic complications,
* a history of previous injury or surgery to the fractured level,
* inability to complete the questionnaires about pain and disability.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Joong Kim, MD, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Derived] Kim HJ, Yi JM, Cho HG, Chang BS, Lee CK, Kim JH, Yeom JS. Comparative study of the treatment outcomes of osteoporotic compression fractures without neurologic injury using a rigid brace, a soft brace, and no brace: a prospective randomized controlled non-inferiority trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1959-66. doi: 10.2106/JBJS.N.00187. PMID 25471910

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Started | 20 | 20 | 20
Completed | 17 | 15 | 17
Not Completed | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Rigid Brace Group: Patients in the rigid brace immobilization group were strictly maintained on bed rest until fitted a thoraco-lumbo-sacral orthosis. Brace is required to be worn at all times except when lying. All patients were instructed to wear the rigid brace for a total of 8 weeks.
  Rigid brace: In rigid brace group, brace is required to be worn at all times except when lying. All patients were instructed to wear the rigid brace for a total of 8 weeks. Then, weaning period requires additional 4 weeks.
- Soft Brace Group: Because soft back brace was a custom-made, it began to be worn when enrollment for the study. Brace is required to be worn at all times except when lying. All patients were instructed to wear the soft brace for a total of 8 weeks.
  Soft brace: In soft brace group, brace is required to be worn at all times except when lying. All patients were instructed to wear the soft brace for a total of 8 weeks. Then, weaning period requires additional 4 weeks.
- Total: Total of all reporting groups
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.25 (10.40) | 66.75 (11.00) | 71.75 (7.96) | 70.25 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 14 | 41
  Male | 7 | 6 | 6 | 19
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index (ODI) at 12 Weeks
Description: The primary outcome was the score for Oswestry Disability Index (ODI) at 12 weeks after compression fracture. The ODI is a self-reported questionnaire measuring back-specific function including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. The questionnaire consists of 10 items each with 6 response levels. Each item is scored from 0 to 5, and the total score is converted to a 0 to 100 scale (zero is equated with no disability and 100 is the maximum disability possible).
Time Frame: 12 weeks after injury
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 35.95 [25.42 to 46.47] | 33.54 [23.79 to 43.29] | 37.83 [26.77 to 48.90]

2. Secondary Outcome: Visual Analog Pain Scale (VAS) for Back Pain
Description: The VAS for back pain comprised a 10-cm line with "none" (0) on one end and "disabled pain" (10) on the other. Participants were asked to place a mark on the 10-cm line, which represented his or her perceived level of back pain, and the measured distance (cm) from the mark to the zero point was considered the score.
Time Frame: 2 weeks, 6 weeks, 12 weeks after injury
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  2 weeks after injury | 5.9 (1.9) | 5.5 (1.8) | 6.8 (1.7)
  6 weeks after injury | 4.6 (2.0) | 5.2 (1.8) | 6.3 (2.0)
  12 weeks after injury | 4.9 (2.0) | 3.4 (2.1) | 4.2 (1.9)

3. Secondary Outcome: Oswestry Disability Index (ODI)
Description: The ODI is a self-reported questionnaire measuring back-specific function including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling. The questionnaire consists of 10 items each with 6 response levels. Each item is scored from 0 to 5, and the total score is converted to a 0 to 100 scale (zero is equated with no disability and 100 is the maximum disability possible).
Time Frame: at 2 weeks, 6 weeks, and 12 weeks after compression fracture.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  2 weeks after injury | 56.84 (17.06) | 53.32 (13.56) | 64.19 (16.12)
  6 weeks after injury | 47.05 (16.22) | 52.53 (14.52) | 57.62 (16.53)
  12 weeks after injury | 42.12 (16.12) | 38.73 (13.78) | 44.25 (17.12)

4. Secondary Outcome: General Health Status
Description: The general health status was assessed with use of the Short Form-36 Health Survey (SF-36) at the initial enrollment and 12 weeks after compression fracture.The raw scores for the eight subscales and the two summaries of the SF-36 (Physical Function,Role Physical, Bodily Pain, General Health, Vitality, Social Function, Role Emotion, and Mental Health, as well as the Physical Component Summary [PCS] and the Mental Component Summary [MCS]) were transformed into norm-based 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability, and the higher the score the less disability. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: at the initial enrollment and 12 weeks after compression fracture
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  SF-36 PCS at the initial enrollment | 29.70 (13.55) | 34.18 (14.58) | 29.87 (11.87)
  SF-36 PCS at 12 weeks after injury | 31.15 (12.45) | 32.75 (14.23) | 33.53 (11.52)
  SF-36 MCS at the initial enrollment | 41.79 (10.31) | 48.29 (14.93) | 42.21 (11.75)
  SF-36 MCS at 12 weeks after injury | 36.53 (11.64) | 37.85 (14.62) | 34.63 (12.43)

5. Secondary Outcome: the Progression of Body Compression Ratio Over All Follow-up Assessments
Description: The anterior body compression ratio was assessed by calculating the ratio between the vertical height of the most compressed anterior section of the injured vertebral body and the posterior vertebral body height at that level
Time Frame: 2 weeks, 6 weeks, and 12 weeks after compression fracture
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Number analyzed (Participants) | 20 | 20 | 20
ratio
  2 weeks after injury | 0.62 (0.05) | 0.67 (0.03) | 0.70 (0.05)
  6 weeks after injury | 0.58 (0.04) | 0.66 (0.04) | 0.65 (0.03)
  12 weeks after injury | 0.57 (0.05) | 0.63 (0.03) | 0.64 (0.03)

ADVERSE EVENTS:
Arm/Group | No Brace Group | Rigid Brace Group | Soft Brace Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Brace Group (N=20) | Rigid Brace Group (N=20) | Soft Brace Group (N=20)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No